CLINICAL TRIAL: NCT07307950
Title: "Healthcare APPlication for Children and Young People With Neuromotor Disabilities": a Digital Tool to Promote Integrated Pediatric Rehabilitation Care for Children and Young People With Disabilities and Their Families: a Mixed-methods Usability-acceptability-impact Study (HAPPY)
Acronym: HAPPY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Principal Investigator, Marietta KERSALE, OT, MSc, PhD student, University Hospital, Brest
Other Study IDs: 29BRC25.0043 - HAPPY
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Children and Adolescents With Neuromotor Impairment; Children and Youth With Special Healthcare Needs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of children followed-up in rehabilitation: Group of 20 children living with neuromotor impairments followed-up in paediatric rehabilitation, with their parents and at least 2 rehabilitation professional per child.

SUMMARY:
The goal of this observational multicentric mixed methods study is to evaluate if the digital application "Deneo Kid", co-designed in France with adolescents, families, rehabilitation providers and researchers, can improve the coordination and quality of rehabilitation care for children and young people with neuromotor disabilities. The main questions it aims to answer are whether the application is easy to use for children, their families, and rehabilitation professionals, is acceptable, whether it helps families and professionals provide more integrated, including more family-centered and coordinated care, and whether it affects communication, relationships, and time and costs related to care coordination.

Rehabilitation providers, families and adolescents ≥ 16 years old will use the "Deneo Kid" secured application for 3 months to share information, track care goals, and communicate with the rehabilitation care team. They will complete short surveys before and after using the application to report on usability, acceptability, quality, and the impact on rehabilitation care. Participants will also take part in interviews or focus groups to share their experiences with the application.

The study will include 20 children, adolescents and young people aged 2 to 25 years living with neuromotor disabilities, followed-up in rehabilitation, their parents or legal guardians, and at least two rehabilitation professionals per child. Four rehabilitation centers in France will participate to the study. Researchers will observe how the application is used in these different rehabilitation settings and collect information on usability, care coordination, user experience, and the time and cost involved in managing care. The results will help determine whether "Deneo Kid" could support better coordination and family-centered rehabilitation for children and young people with disabilities and provide a foundation for larger future studies, to evaluate the effectiveness of the application.

DETAILED DESCRIPTION:
Context Chronic diseases are increasing, and healthcare is becoming more complex. Integrated care-that is, care that is coordinated, person-centered, and continuous-is essential to improve efficiency. In pediatric rehabilitation, coordination between the child, their family, and professionals working in hospitals, rehabilitation centers, integrated healthcare and social settings, outpatient settings, private practice is particularly critical. Effective coordination helps promote the child's participation in all areas of life and supports them through major life transitions, such as starting school or moving from adolescence to adulthood.

In this context, the digital application "Deneo Kid" was developed at the University Hospital of Brest through a partnership between the company Deneo, which already developed a shared portal for adult sports rehabilitation, and the BEaCHILD research team, specialized in child disability. It was designed based on qualitative studies exploring the needs of parents of children with disabilities (PitchRehab, supported by the Ildys Foundation), young people with disabilities (KidChildRehab, supported by the University Hospital of Brest), and professionals in rehabilitation, education, and leisure (ProChildRehab, supported by the University Hospital of Brest). "Deneo Kid" aims to connect children, their families, and rehabilitation professionals around a coordinated care and life plan centered on their needs, in order to promote integrated pediatric rehabilitation using a digital tool.

Funding from the Fondation de l'Avenir has been obtained to conduct a usability and impact study of the application. Additional funding has been requested from IReSP to explore the social determinants of adoption and the economic impact of the application with the support of a sociologist and a health economist from IMT Atlantique, as part of the same usability study.

To achieve this, the "Deneo Kid" application will be tested for 3 months with a cohort of users composed of 20 "teams," each including one child living with a neuromotor disability (cerebral palsy, neuromuscular disease, neurodevelopmental disease with motor impairments, etc.), their parents/legal guardians, and at least two rehabilitation professionals involved in their rehabilitation. Participants will be recruited from four pediatric rehabilitation centers in France. A mixed-methods approach will be used, including quantitative data collection and analysis (pre- and post-intervention questionnaires for users, anonymized application usage data collected via Deneo, and costs associated with coordination with and without the application) and qualitative data collection and analysis (interviews and focus groups before and after the study, digital journals, and direct observations).

This first small-scale experimental study will provide a better understanding of the usability, acceptability and impact of "Deneo Kid" across different pediatric rehabilitation settings and the factors contributing to its success. It will also provide a solid foundation for future larger-scale studies, contributing to improvements in the quality and efficiency of pediatric rehabilitation care.

Target Population The end users of the "Deneo Kid" digital solution include children and young people with disabilities aged 0-25 years, parents or legal guardians of these children, and rehabilitation professionals such as physicians, physiotherapists, occupational therapists, psychomotor therapists, psychologists, speech therapists, specialized educators, and adapted physical activity educators. The term "parents or family" is used throughout the text for simplicity but includes legal guardians.

Primary Objective The primary objective of this study is to evaluate the usability of the "Deneo Kid" application among the described user cohort.

Secondary Objectives

The secondary objectives of the study are:

1. To evaluate the use of the "Deneo Kid" application by all participants.
2. To assess the quality of the application from the perspective of all users.
3. To evaluate the impact of the application on the provision of integrated care from the perspective of families.
4. To assess the effect of the application on the implementation of family-centered care from the perspectives of both families and professionals.
5. To evaluate the acceptability of the application from the viewpoint of all participants.
6. To analyze the influence of the application on communication and relational dynamics among stakeholders.
7. To identify social determinants that affect the adoption of the application in different contexts.
8. To compare the time and costs of care coordination before and after using the application from the perspectives of families and professionals.

Primary Outcome Measure The primary outcome is usability, assessed using the System Usability Scale (SUS), completed by adolescents over 16, their parents, and the rehabilitation professionals who follow them.

Secondary Outcome Measures

1. Application use: Usage will be monitored through anonymized back-office data, including login times, average connection durations, and feature usage over the three months.
2. Application quality: Quality will be assessed using the validated Mobile Application Rating Scale (MARS) for young adults, families, and professionals after three months of use.
3. Integrated care: Families will complete the Pediatric Integrated Care Survey (PICS) before and after three months to evaluate the impact on integrated care.
4. Family-centered care: Families will complete the Measure of Processes of Care (MPOC) questionnaires, and professionals will complete the MPOC-Service Providers (MPOC-SP) questionnaire before and after three months to assess family-centered care practices.
5. Acceptability: Acceptability will be evaluated through the questionnaire Theoretical Framework Acceptability and through interviews or focus groups with adolescents, parents, and professionals conducted in person or via videoconference.
6. Relational dynamics and communication: interviews and observations on site will assess communication and relationships among participants.
7. Social determinants of adoption: Socio-demographic data collected before the study will be analyzed to identify factors affecting adoption.
8. Time and coordination costs: Direct costs (Deneo subscription) and indirect costs (time spent using the application) will be collected via application usage statistics and coordination practice questionnaires before and after the study.

Methodology This is a multicenter, prospective observational study evaluating professional practices using a mixed-methods design with quantitative and qualitative data across 20 child-family-professional teams.

Statistics Each participant will be assigned a pseudonym, and only the principal investigators will have access to the key linking names to pseudonyms. Quantitative data will be stored on a secure server in Excel files and analyzed descriptively, reporting frequencies, means with standard deviations, or medians with interquartile ranges depending on the data type. The primary criterion of usability considers a mean SUS score above 51 as acceptable.

Qualitative data from interviews and focus groups will be recorded using Zebrix, a local secure platform of the university hospital of Brest, and transcribed verbatim using AI. Analysis will follow the six-phase thematic analysis method of Braun & Clarke (2016) using NVivo14 software.

Inclusion Criteria Children and young people aged 0-25 with a physical disability (such as acquired brain injury, musculoskeletal disorders, rare diseases, congenital heart conditions) causing participation limitations according to the International Classification of Functioning, Disability and Health (WHO, 2007), who are followed in rehabilitation at least once per week by at least two professionals in different sectors with the goal of promoting autonomy and participation. Parents or legal guardians must have access to a computer, smartphone, or tablet. Rehabilitation professionals must work with children with disabilities and have access to digital devices.

Exclusion Criteria Refusal to participate.

Number of Participants The study aims to include 20 children/young people, their parents, and at least two rehabilitation professionals per child. The total number of participants using the application for three months is expected to be between 80 and 100.

Timeline Enrollment will take place over 12 months. Each participant will use the application for three months, between November 2025 and June 2026. The total study duration, including enrollment and follow-up, is 12 months, with data collection and processing expected to take 18 months.

ELIGIBILITY:
Inclusion Criteria for children:

* Aged 2 to 25 years.
* Presenting a neuromotor impairment (such as cerebral palsy, acquired brain injury, musculoskeletal disorders, rare diseases, congenital heart conditions,...) that results in limitations in participation, according to the International Classification of Functioning, Disability and Health (ICF, WHO 2007).
* Receiving rehabilitation at least once per week from at least two professionals in different care settings (e.g., healthcare, integrated health and social care, and outpatient settings) with a focus on promoting autonomy and participation.

Inclusion criteria for parents:

* Being the parent or legal guardian of a child meeting the criteria above.
* Having access to a computer, smartphone, or tablet.

Inclusion criteria for rehabilitation professionals:

* Working with children with disabilities in pediatric rehabilitation (including physicians, physiotherapists, occupational therapists, psychomotor therapists, psychologists, speech therapists, specialized educators, or adapted physical activity educators).
* Practicing in healthcare, integrated health and social care, or outpatient/private practice settings.
* having access to a computer, smartphone, or tablet.

Exclusion Criteria:

* Refusal to participate.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with neuromotor impairments followed up in four paediatric rehabilitation settings in France: healthcare, integrated health and social care, and outpatient/private practice settings.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the app | from enrollment (beginning of use of the app) to the end of the application test at 3 months
  Usability of the "Deneo Kid" application from the perspective of all end-users (adolescents, families, professionals)

SECONDARY OUTCOMES:
Acceptability | From enrollment (beginning of the use of the app) to the end of the use of the app at 3 months
  Acceptability of the "Deneo Kid" application from the viewpoint of all end-users (adolescents and young people, families, professionals)
Impact on integrated care | From enrollment (beginning of the use of the app) to the end of the use of the app at 3 months
  The impact of the "Deneo Kid" application on the provision of integrated care from the viewpoint of families (PICS, MPOC), professionals (MPOC-SP), and adolescents (interviews/focus groups).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Result] Cornec G, Drewnowski G, Desguerre I, Toullet P, Boivin J, Bodoria M, De La Cruz J, Brochard S; ESPaCe group. Determinants of satisfaction with motor rehabilitation in people with cerebral palsy: A national survey in France (ESPaCe). Ann Phys Rehabil Med. 2021 May;64(3):101314. doi: 10.1016/j.rehab.2019.09.002. Epub 2019 Oct 3. PMID 31586683
- [Result] Ziniel SI, Rosenberg HN, Bach AM, Singer SJ, Antonelli RC. Validation of a Parent-Reported Experience Measure of Integrated Care. Pediatrics. 2016 Dec;138(6):e20160676. doi: 10.1542/peds.2016-0676. PMID 27940672
- [Result] Cassidy L, Quirke MB, Alexander D, Greene J, Hill K, Connolly M, Brenner M. Integrated care for children living with complex care needs: an evolutionary concept analysis. Eur J Pediatr. 2023 Apr;182(4):1517-1532. doi: 10.1007/s00431-023-04851-2. Epub 2023 Feb 13. PMID 36780041
- [Result] Rosenbaum P, Gorter JW. The 'F-words' in childhood disability: I swear this is how we should think! Child Care Health Dev. 2012 Jul;38(4):457-63. doi: 10.1111/j.1365-2214.2011.01338.x. Epub 2011 Nov 1. PMID 22040377
- See also: Related Info — https://beachild.fr/
- See also: Related Info — https://deneo.fr/